CLINICAL TRIAL: NCT02297659
Title: Use of Hypertonic Saline After Damage Control Laparotomy to Improve Early Primary Fascial Closure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Antonio Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Valerie Sams, Acute Care Surgery Fellow, San Antonio Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 397284-1
Record Dates: First submitted 2014-08-01; First posted 2014-11-21 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Open Abdomen After Damage Control Laparotomy
Keywords: damage control; resuscitation; laparotomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Crystalloid resuscitation (Active Comparator): Patients to receive normal saline resuscitation at a rate of 30cc/hr.
  Interventions: Procedure: Primary Fascial Closure; Device: wound vac dressing application
- Hypertonic saline resuscitation (Active Comparator): Patients to receive 3% hypertonic saline resuscitation at a rate of 30cc/hr.
  Interventions: Procedure: Primary Fascial Closure; Device: wound vac dressing application

INTERVENTIONS:
Procedure: Primary Fascial Closure — Abdominal wall closure following damage control laparotomy.
Device: wound vac dressing application — temporary abdominal wall closure with this device after damage control laparotomy
  Other Names: AbThera woulnd vac (KCI)

SUMMARY:
Damage control laparotomy (DCL) has proven to be a successful means to improve survival in severely injured patients.1-5 However, the consequences of not being able to close the fascia after the initial operation due to significant resuscitation leading to bowel and retroperitoneal edema, abdominal compartment syndrome, and continued acidosis, coagulopathy and hypethermia6-7 has led to a new challenge. Delays in primary fascial closure (PFC) contributes to increased fluid losses and nutritional demands,8-9 abdominal wall hernias, enterocutaneous fistula, and intra-abdominal infections.10-13 Hypertonic saline (HTS) use after DCL has been suggested to reduce bowel edema and resuscitation volumes, thus allowing for a quicker time to closure.14 Investigators will randomize patients to receiving HTS or standard crystalloid solutions after DCL and compare the time to PFC, rate of successful closure, and rate of complications associated with an open abdomen. The current failure rate of PFC after DCL is approximately 25%. Investigators believe they can improve PFC rates using hypertonic saline.

DETAILED DESCRIPTION:
The use of HTS after DCL may decrease the rate of failure to achieve PFC and reduce the number of complications associated with an open abdomen.

Research Questions:

1. Primary Objective: Is there a higher rate of PFC among patients who undergo DCL and temporary abdominal closure when using HTS versus standard crystalloid resuscitation?
2. Secondary Objectives: Does successful and faster PFC reduce ICU, ventilator and hospital days?
3. Does faster and more successful PFC result in lower morbidity to include enterocutaneous fistula (ECF), intra-abdominal abscess (IAA), abdominal wall hernia, and anastomotic failure?

DCL is a common procedure wounded warriors undergo due to blast and other blunt and penetrating mechanisms of injury. This results in a significant population of warriors at risk for all of the complications and comorbidities that accompany an open abdomen. Thus, finding ways to not only achieve PFC but also to decrease the time to PFC will reduce these unwanted events.

The protocol design is a multi-institutional, prospective, double blind, randomized controlled trial of patients who undergo DCL for abdominal trauma requiring temporary abdominal closure and return to operating room for definitive treatment. All participating facilities are Level I Trauma Centers. Currently, the standard of care for damage control resuscitation involves all intravenous fluid solutions utilized in this study; normal saline, Ringer's lactate, Plasmalyte, and 3% saline (HTS). However, the type of fluid is selected based on surgeon preference alone. Investigators will randomize patients to normal saline at a resuscitation rate of 30 cc/hr or to 3% saline (HTS) at a resuscitation rate of 30cc/hr which will be initiated upon arrival to the ICU.

ELIGIBILITY:
Inclusion Criteria:

* All admissions of trauma patients who sustain trauma necessitating damage control laparotomy.
* Male and female patients 18 years or older.

Exclusion Criteria:

* Children (<18 years old), prisoners, or pregnant patients.
* Patients who have more than 1/3 loss of abdominal wall due to trauma.
* Patients with baseline serum sodium of <120 mEq/L or >155 mEq/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who achieve primary fascial closure | 2 weeks
  Is there a higher rate of PFC among patients who undergo DCL and temporary abdominal closure when using HTS versus standard crystalloid resuscitation?

SECONDARY OUTCOMES:
number of ICU free days | 30 days
  Does successful and faster PFC reduce ICU days?
number of enterocutaneous fistula | 90 days
  Does faster and more successful PFC result in reduction enterocutaneous fistula (ECF)?
number of intra abdominal abscess | 90 days
  Does faster and more successful PFC result in reduction of intra-abdominal abscess (IAA)?
number of abdominal wall hernias | 90 days
  Does faster and more successful PFC result in reduction in abdominal wall hernia?
number of anastomotic failure | 90 days
  Does faster and more successful PFC result in a reduction in anastomotic failure?
number of ventilator free days | 30 days
  Does successful and faster PFC reduce ventilator days?
number of hospital free days | 30 days
  Does successful and faster PFC reduce hospital days?

CONTACTS AND LOCATIONS:
Locations (1):
- San Antonio Military Medical Center, San Antonio, Texas, United States

REFERENCES:
- [Background] Harvin JA, Mims MM, Duchesne JC, Cox CS Jr, Wade CE, Holcomb JB, Cotton BA. Chasing 100%: the use of hypertonic saline to improve early, primary fascial closure after damage control laparotomy. J Trauma Acute Care Surg. 2013 Feb;74(2):426-30; discussion 431-2. doi: 10.1097/TA.0b013e31827e2a96. PMID 23354234